CLINICAL TRIAL: NCT06589869
Title: To Investigate the Effect of High-Intensity Focused Electromagnetic (HIFEM) Technology in the Treatment of Stress Urinary Incontinence Compared With Standard of Care in Chinese Men Who Had Undergone Robotic Radical Prostatectomy
Brief Title: Effect of High-Intensity Focused Electromagnetic (HIFEM) Technology in the Treatment of SUI in Chinese Men Undergone Robotic Radical Prostatectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chi Fai NG, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CRE-2021.506-T
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Urinary Incontinence , Stress; Prostatectomy
Keywords: stress urinary incontinence; prostatectomy
MeSH Terms: conditions — Urinary Incontinence, Stress | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Standard of care. Perioperative education for information related to prostatectomy and pelvic floor exercise training. Patient were advice to perform pelvic floor exercise at least 30 times per day
  Interventions: Other: Standard of care
- EM Chair (Experimental): Patients who randomised to intervention group (Arm A) will receive HIFEM assisted (BTL EMsella) pelvic floor muscle training for total 6 sessions (2 session per week, 30 minutes per session with modulated intensity) plus standard of care. The intervention will be started within 2 weeks after Foley Catheter removed. Patients will attend follow up for training and at 1, 3 and 6 month post-operatively.
  Interventions: Device: EM Chair

INTERVENTIONS:
Device: EM Chair — Patients who randomised to intervention group (Arm A) will receive HIFEM assisted (BTL EMsella) pelvic floor muscle training for total 6 sessions (2 session per week, 30 minutes per session with modulated intensity) plus standard of care. The intervention will be started within 2 weeks after Foley Catheter removed. Patients will attend follow up for training and at 1, 3 and 6 month post-operatively.
  Arms: EM Chair
Other: Standard of care — Standard of care. Perioperative education for information related to prostatectomy and pelvic floor exercise training. Patient were advice to perform pelvic floor exercise at least 30 times per day
  Arms: Standard of Care

SUMMARY:
This is a prospective, randomized trial to evaluate the efficacy and safety of High-Intensity Focused Electromagnetic (HIFEM) Technology in the treatment of stress urinary incontinence compared with standard of care in Chinese men who had undergone robotic radical prostatectomy.

DETAILED DESCRIPTION:
This is a prospective randomised control trial of consecutive patients with prostatectomy to have either standard of care versus HIFEM assisted pelvic floor exercise. Randomization will be performed for patients when the subject has completed the informed consent for study participation. Randomization will be performed in 1:1 ratio into 2 arms: HIFEM assisted (BTL EMsella) pelvic floor muscle training (Arm A) plus Standard of care or Standard of care (Arm B).

ELIGIBILITY:
Inclusion Criteria:

* Undergone robotic radical prostatectomy
* Able to carry out 1-hour pad test
* Voluntary participation and signing of the informed consent form

Exclusion Criteria:

* Pre-existing stress urinary incontinence
* Post-void residual urine greater than 200ml
* Active urinary tract infection
* Urethral or bladder fistula
* History of pelvic irradiation
* Neurological condition (Spinal cord problems, stroke with poor neurological recovery, epilepsy, Parkinson disease, multiple sclerosis)
* Previous surgery for SUI
* Concurrent medication with diuretics, serotonin-norepinephrine reuptake inhibitors or any other medication known to worsen incontinence
* Condition contraindicated for electromagnetic therapy i.e. Arrhythmia, on a pacemaker or implanted metallic device; Coagulopathy or on anticoagulant

Min Age: 18 Months | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 184 (Estimated)
Dates: Start 2022-07-29 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Weight of 1-hour pad test | Baseline, Month 1, Month 3 and Month 6
  Weight of 1-hour pad test

SECONDARY OUTCOMES:
Severity of Incontinence. | Baseline, Month 1, Month 3 and Month 6
  It is evaluated by International Consultation on Incontinence Questionnaire-Urinary Incontinence Short FormInternational Consultation on Incontinence Questionnaire-Urinary Incontinence Short Form. The ICIQ score with a range from 0-21; the higher the score the worse of incontinence
Sexual Function | Baseline, Month 1, Month 3 and Month 6
  It is evaluated by International Index of Erectile Function Score (IIEF-5). The IIEF-5 score is the sum of the ordinal response to the 5 items. The lowest the score, the more severe of erectile dysfunction
Severity of Incontinence | Baseline, Month 1, Month 3 and Month 6
  The number of pads used
Complications | Month 1, Month 3 and Month 6
  It is evaluated by CTCAE Grade 5

CONTACTS AND LOCATIONS:
Overall Officials: Chi Fai NG, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

REFERENCES:
- [Background] Anderson CA, Omar MI, Campbell SE, Hunter KF, Cody JD, Glazener CM. Conservative management for postprostatectomy urinary incontinence. Cochrane Database Syst Rev. 2015 Jan 20;1(1):CD001843. doi: 10.1002/14651858.CD001843.pub5. PMID 25602133
- [Background] Kashanian M, Ali SS, Nazemi M, Bahasadri S. Evaluation of the effect of pelvic floor muscle training (PFMT or Kegel exercise) and assisted pelvic floor muscle training (APFMT) by a resistance device (Kegelmaster device) on the urinary incontinence in women: a randomized trial. Eur J Obstet Gynecol Reprod Biol. 2011 Nov;159(1):218-23. doi: 10.1016/j.ejogrb.2011.06.037. Epub 2011 Jul 7. PMID 21741151
- [Background] Fernandez RA, Garcia-Hermoso A, Solera-Martinez M, Correa MT, Morales AF, Martinez-Vizcaino V. Improvement of continence rate with pelvic floor muscle training post-prostatectomy: a meta-analysis of randomized controlled trials. Urol Int. 2015;94(2):125-32. doi: 10.1159/000368618. PMID 25427689
- [Background] Samuels JB, Pezzella A, Berenholz J, Alinsod R. Safety and Efficacy of a Non-Invasive High-Intensity Focused Electromagnetic Field (HIFEM) Device for Treatment of Urinary Incontinence and Enhancement of Quality of Life. Lasers Surg Med. 2019 Nov;51(9):760-766. doi: 10.1002/lsm.23106. Epub 2019 Jun 7. PMID 31172580
- [Background] Sanda MG, Dunn RL, Michalski J, Sandler HM, Northouse L, Hembroff L, Lin X, Greenfield TK, Litwin MS, Saigal CS, Mahadevan A, Klein E, Kibel A, Pisters LL, Kuban D, Kaplan I, Wood D, Ciezki J, Shah N, Wei JT. Quality of life and satisfaction with outcome among prostate-cancer survivors. N Engl J Med. 2008 Mar 20;358(12):1250-61. doi: 10.1056/NEJMoa074311. PMID 18354103
- [Background] Wang W, Huang QM, Liu FP, Mao QQ. Effectiveness of preoperative pelvic floor muscle training for urinary incontinence after radical prostatectomy: a meta-analysis. BMC Urol. 2014 Dec 16;14:99. doi: 10.1186/1471-2490-14-99. PMID 25515968
- [Background] Wilt TJ, Brawer MK, Jones KM, Barry MJ, Aronson WJ, Fox S, Gingrich JR, Wei JT, Gilhooly P, Grob BM, Nsouli I, Iyer P, Cartagena R, Snider G, Roehrborn C, Sharifi R, Blank W, Pandya P, Andriole GL, Culkin D, Wheeler T; Prostate Cancer Intervention versus Observation Trial (PIVOT) Study Group. Radical prostatectomy versus observation for localized prostate cancer. N Engl J Med. 2012 Jul 19;367(3):203-13. doi: 10.1056/NEJMoa1113162. PMID 22808955